CLINICAL TRIAL: NCT03784157
Title: Study Of The Metabolic Parameters Of Uterine Muscle Cells In Cold Ischemia From Hysterectomies Programmed For Benign
Brief Title: Study Of The Metabolic Parameters Of Uterine Muscle Cells
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7222
Record Dates: First submitted 2018-12-13; First posted 2018-12-21 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2018-12

CONDITIONS: Ischemia
Keywords: Hysterotomy; UTERINE MUSCLE CELLS; ISCHEMIA; COLD ISCHEMIA
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, no transplant has allowed pregnancy from a donor in a state of brain death. One of the main reservations lies in the ischemic properties of the uterine graft between the sampling time and the grafting time.

Investigators propose to carry out a prospective monocentric study at the University Hospitals of Strasbourg in 2018/2019: the objective would be to study physiologically the time of ischemia of the uterine muscle The objective is to carry out a preparatory study on healthy uteri to study the ischemic properties of uterine muscle from living markers: study of mitochondrial respiration and free radical production on uterine muscle samples If the markers are reliable, they would then be used to measure the ischemia of whole uteri collected at the end of the multi-organ retrieval process from donors in a state of brain death and stored in tissue survival media.

ELIGIBILITY:
Inclusion criteria:

* - Adult patient
* Patient benefiting from the routine management of a programmed hysterectomy by vaginal, laparoscopic or laparotomy for benign pathologies (fibroma, adenomyosis, genital prolapse,...) within the CMCO
* Patient consenting to the use of cells from her uterus for incineration for research purposes
* Patient giving her consent for the use of her medical data for the purposes of this research.
* Patient agreeing to participate in the study

Exclusion criteria:

* - Patient refusing to participate in the study
* Patient under the protection of justice
* Patient under guardianship or curatorship
* Suspicion of gynaecological malignant pathology
* Pregnant or breastfeeding woman
* Impossibility to give the subject informed information (difficulties in understanding the subject...)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient benefiting from the routine management of a programmed hysterectomy by vaginal, laparoscopic or laparotomy for benign pathologies
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
Ischemia | 1 hour after sampling
  Study physiologically the time of ischemia of the uterine muscle 1 hour after sampling

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GARBIN, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Gynécologie - CMCO, Strasbourg, France